CLINICAL TRIAL: NCT07034963
Title: Study on the Effective Dose and Safety of Esketamine in Hysteroscopic Surgery Under Monitored Anesthesia Care
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Lijuan Yan, Scientific Research Secretary of the Anesthesiology Department, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: XMFHIIT-2025SL092
Record Dates: First submitted 2025-05-29; First posted 2025-06-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Intrauterine Polyp; Intrauterine Synechiae
Keywords: ambulatory hysteroscopic surgery; monitored anesthesia care; esketamine; cervical dilation response; Intrauterine lesion
MeSH Terms: conditions — Gynatresia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This research will be divided into two stages. (i) In Phase one, a prospective dose discovery study using the Dixon sequential method will be conducted, aiming to determine the median effective dose (ED50) and 95% effective dose (ED95) of esketamine in inhibiting cervical response. The test will continue until six cross-pairings are obtained. The sample size is approximately 33. (ii) The investigators will conduct a single-center, randomized, double-blind controlled trial in Phase Two to evaluate the safety of the esketamine ED95 dose under the monitoring anesthesia care program based on the incidence of respiratory depression. The intervention group will be injected with the dose of esketamine ED95; the control group will be injected with remifentanil 1μg∙kg-1. Both groups of patients will receive the same sedation regimen. The sample size is approximately 62.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Determine the ED50 and ED95 of esketamine by Dixon's up-and-down method (Experimental): According to Dixon's up-and-down sequential design, esketamine will be initiated at 0.3 mg∙kg-1 intravenously, followed by dose adjustments (0.02 mg∙kg-1 increments/decrements) based on somatic responses to cervical dilation (positive: any movement; negative: no movement). The tests will continue until six crossover pairs are achieved.
  Interventions: Drug: Determine the ED50 and ED95 of esketamine
- Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression (Active Comparator): The intervention group will be injected with the dose of esketamine ED95; the control group will be injected with remifentanil 1μg∙kg-1. Both groups of patients will receive the same Monitoring Anesthesia Care (MAC) regimen, namely, remifentanil will be continuously pumped at a rate of 5μg∙kg∙h-1 combined with dexmedetomidine (a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance dose of 0.4 μg∙kg-1∙h-1). Intravenous injection of 100 mg of flurbiprofen axetil for auxiliary analgesia. Intravenous injection of 4 mg of ondansetron to prevent nausea and vomiting. The study at this stage will evaluate the safety of the dose of esketamine ED95 through the incidence of respiratory depression.
  Interventions: Drug: Intravenous the dose of esketamine ED95; Drug: Intravenous remifentanil 1μg∙kg-1

INTERVENTIONS:
Drug: Determine the ED50 and ED95 of esketamine — According to Dixon's up-and-down sequential design, esketamine will be initiated at 0.3 mg∙kg-1 intravenously, followed by dose adjustments (0.02 mg∙kg-1 increments/decrements) based on somatic responses to cervical dilation (positive: any movement; negative: no movement). The tests will continued until six crossover pairs are achieved.
  Other Names: Remifentanil will be continuously pumped at a rate of 5μg∙kg∙h-1 combined with dexmedetomidine (a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance dose of 0.4 μg∙kg-1∙h-1).
  Arms: Determine the ED50 and ED95 of esketamine by Dixon's up-and-down method
Drug: Intravenous the dose of esketamine ED95 — The intervention group will be injected with the dose of esketamine ED95.
  Other Names: Remifentanil will be continuously pumped at a rate of 5μg∙kg∙h-1 combined with dexmedetomidine (a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance dose of 0.4 μg∙kg-1∙h-1).
  Arms: Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression
Drug: Intravenous remifentanil 1μg∙kg-1 — The control group will be injected with remifentanil 1μg∙kg-1.
  Other Names: Remifentanil will be continuously pumped at a rate of 5μg∙kg∙h-1 combined with dexmedetomidine (a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance dose of 0.4 μg∙kg-1∙h-1).
  Arms: Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression

SUMMARY:
Cervical dilation-induced somatic responses remain a critical challenge in ambulatory hysteroscopic surgery. Esketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, exhibits unique analgesic and sedative properties that may enhance perioperative somatic response inhibition. However, the effective dose of esketamine under dexmedetomidine-remifentanil based monitored anesthesia care (MAC) during ambulatory hysteroscopic surgery remains to be determined. This prospective dose-finding study aimed to establish the median effective dose (ED50) and 95% effective dose (ED95) of esketamine for cervical response suppression. Afterwards, the investigators will conduct an RCT study to evaluate the safety of the dose of esketamine ED95 through the incidence of respiratory depression.

DETAILED DESCRIPTION:
This research will be divided into two stages. (i) In Phase one, a prospective dose discovery study using the Dixon sequential method will be conducted, aiming to determine the median effective dose (ED50) and 95% effective dose (ED95) of esketamine in inhibiting cervical response. Esketamine will be initiated by intravenous infusion at 0.3 mg∙kg-1, followed by somatic response based on cervical dilation (positive: any exercise; negative: no movement). Dose adjustment will be carried out, with a dose fluctuation step of 0.02 mg∙kg-1 up and down. All patients will receive a standardized anesthesia regimen, including continuous infusion of remifentanil at a dose of 5 μg∙kg∙h-1, combined with dexmedetomidine (infusion at a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance infusion at 0.4 μg∙kg-1∙h-1). The test will continue until six cross-pairings are obtained. Probabilistic regression analysis will be used to calculate the ED50 and ED95 of esketamine with a 95% confidence interval.

(ii) The investigators will conduct a single-center, randomized, double-blind controlled trial in Phase Two to evaluate the safety of the esketamine ED95 dose under the monitoring anesthesia care program based on the incidence of respiratory depression. The intervention group will be injected with the dose of esketamine ED95; the control group will be injected with remifentanil 1μg∙kg-1. Both groups of patients will receive the same sedation regimen, namely remifentanil will be continuously pumped at a rate of 5μg∙kg∙h-1 combined with dexmedetomidine (pumped at a loading dose of 0.6 μg∙kg-1 for 10 minutes, followed by maintenance pumping at 0.4 μg∙kg-1∙h-1). Intravenous injection of 100 mg of flurbiprofen axetil for auxiliary analgesia. Intravenous injection of 4 mg of ondansetron to prevent nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 55 years;
* ASA physical status Ⅰ or Ⅱ;
* Body mass index (BMI) 18 - 28 kg∙m-2;
* Scheduled for elective diagnostic/therapeutic hysteroscopy.

Exclusion Criteria:

(i) Pharmacological contraindications:

* Known hypersensitivity to study medications (esketamine, remifentanil, dexmedetomidine);
* Opioid or benzodiazepine medications dependence;
* Analgesic/psychotropic medication use within 48 hours preoperatively;
* Participation in any other drug clinical trial within the preceding three months.

(ii) Comorbidities:

* Significant cardiopulmonary dysfunction (NYHA III-IV, FEV₁/FVC <70%);
* Hepatic impairment (Child-Pugh B/C);
* Uncontrolled hypertension, intracranial hypertension, intraocular hypertension or hyperthyroidism;
* Neurological/psychiatric conditions (epilepsy, schizophrenia, depression);
* Active gastroesophageal reflux disease (GERD-Q score ≥8). (iii) Airway/Perioperative Risks:
* Anticipated difficult airway (Mallampati III-IV, thyromental distance <6 cm) or airway stenosis;
* Non-fasted status (solids <8h, clear fluids <2h preoperatively).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cervical dilation-induced somatic responses | Day 1 (During the surgery at the first stage of the research)
  Positive: Body movement or complaint of pain. Negative: No body movement or no reported pain. This scale will be administered during the surgery at the first stage of the research.
Incidence of respiratory depression | Day 1 (T2-T6 of the second stage of the research)
  The primary outcome is the incidence of respiratory depression, which is defined as SpO2 <90% or EtCO2 >55 mmHg.
  By comparing with the control group, evaluate the safety of ED95 of esketamine by the incidence of respiratory depression at T2-T6 of the second stage of the research.
  T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.

SECONDARY OUTCOMES:
HR | Day 1 (T1-T6 of the first and second stages of the research)
  HR: heart rate. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.
MAP | Day 1 (T1-T6 of the first and second stages of the research)
  MAP: Mean Arterial Pressure. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.
RR | Day 1 (T1-T6 of the first and second stages of the research)
  RR: respiratory rate. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.
SPO2 | Day 1 (T1-T6 of the first and second stages of the research)
  SPO2: peripheral oxygen saturation. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.
EtCO2 | Day 1 (T2-T6 of the first and second stages of the research)
  EtCO2: End-expiratory carbon dioxide. SPO2: peripheral oxygen saturation. T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU.
Adverse events | Day 1 (T2-T9 of the first and second stages of the research)
  Adverse events will encompass a range of systems, including the cardiovascular system (eg. high/low blood pressure and sinus tachycardia/bradycardia), as well as symptoms such as nausea, vomiting, dizziness, and mental symptoms.
  T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations; T6: In the PACU. T7 to T9: 2, 6, and 24 hours after the procedure.
NRS | Day 1 (T7-T9 of the first and second stages of the research)
  The Numeric Rating Scale (NRS) will be utilized to assess postoperative pain, with a range of 0 representing no pain and 10 representing severe pain. This scale will be administered at 2, 6, and 24 hours following the procedure.
  T7 to T9: 2, 6, and 24 hours after the procedure.
The need for remedial analgesia | Day 1 (T7-T9 of the first and second stages of the research)
  The consumption of remedial analgesia will be the total consumption of acetaminophen documented at 2, 6, and 24 hours after the procedure.
  T7 to T9: 2, 6, and 24 hours after the procedure.
Induction duration | Day 1 of the first and second stages of the research
  Induction duration is defined as the period from the start of anaesthetic drug injection to the commencement of the surgical procedure at the first and second stages of the research.
Duration of awakening | Day 1 of the first and second stages of the research
  Duration of awakening is defined as the period from the conclusion of the surgical procedure to the moment of eye-opening.
PACU time | Day 1 of the first and second stages of the research
  The time from patient admission to the PACU until the fulfillment of the criteria for PACU discharge.
Discharge time | Day 1 of the first and second stages of the research
  The interval between patient admission to the operating room and the fulfillment of the criteria for hospital discharge.
Success rate of anesthesia | Day 1 (T2-T5 of the second stage of the research)
  Anesthesia success will be defined as inadequate analgesia requiring ≤3 rescue doses of remifentanil within 10 min throughout the procedure. The success rate of anesthesia will be calculated by dividing the number of successful anesthesia cases by the total number of cases.
  T2: 60 seconds after esketamine injection; T3: During vaginal disinfection; T4: During cervical dilation; T5: During intrauterine operations.
The satisfaction of gynecologists | Day 1 of the second stage of the research
  The satisfaction score of gynecologists will be collected postoperatively on Day 1, using a scale ranging from 0 to 10, with 0 representing dissatisfaction and 10 representing very satisfied.
The satisfaction of patients | Day 2 of the second stage of the research
  The satisfaction of patients will be collected postoperatively on Day 2, using a scale ranging from 0 to 10, with 0 representing dissatisfaction and 10 representing very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Yan, Principal Investigator — Department of Anesthesiology, The First Affiliated Hospital of Xiamen University
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital of Xiamen University, 55 Zhenhai Road, Xiamen, China, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan L, Wang X, Wei J, Zhang M, Yang B. Prospective Dose-Finding of Esketamine for Suppressing Cervical Dilation Response in Ambulatory Hysteroscopy Under Monitored Anesthesia Care. Drug Des Devel Ther. 2025 Dec 7;19:10835-10845. doi: 10.2147/DDDT.S557340. eCollection 2025. PMID 41393327